CLINICAL TRIAL: NCT01587443
Title: A Comparison of Patient-Reported, Economic and Clinical Outcomes Between Hemodialysis and Peritoneal Dialysis Patients in a Multi-Ethnic Asian Population
Brief Title: Comparison of Outcomes Between Hemodialysis and Peritoneal Dialysis Patients in a Multi-Ethnic Asian Population
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Priscilla How, Pharm.D., BCPS, Assistant Professor, National University of Singapore
Other Study IDs: DSRB Domain E/2011/02160
Record Dates: First submitted 2012-04-26; First posted 2012-04-30 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Stage 5 Chronic Kidney Disease; Hemodialysis; Peritoneal Dialysis
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Hemodialysis
- Peritoneal dialysis

SUMMARY:
End-stage renal disease (ESRD) presents a heavy burden on a patient's psychological and social life, as well as overall quality of life (QoL). Health-related quality of life (HRQoL) in dialysis patients measures the physical, social or emotional well-being that is affected by ESRD and/or its treatment, and has been increasingly used as an outcome measure in interventional studies. Additionally, associations between social support and QoL have been observed, indicating that improved social support could improve HRQoL, morbidity and mortality in ESRD patients. However, it is not clear if hemodialysis (HD) and peritoneal dialysis (PD) have different impacts on HRQoL. Furthermore, comparisons of HRQoL and social support between HD and PD patients in the multiethnic society of Singapore have not been evaluated. As such, the investigators propose to conduct this cross-sectional study in the investigators local multiethnic ESRD patient population to evaluate and compare patient-reported outcomes (HRQoL and social support), economic and clinical laboratory outcomes in HD and PD patients.

All chronic HD and PD patients seen in NUH outpatient renal or PD clinic will be included in this cross-sectional, observational study. Information on patient demographics, medical/medication histories, dialysis vintage, clinical laboratory data and associated medical costs will be obtained from clinic notes, electronic medical records and hospital databases. Patient-reported outcomes will be determined from scores of the Kidney Disease Quality of Life-Short Form, EuroQol 5 Dimensions, Family Functioning Measure, Oslo-3 Social Support Scale, Multidimensional Scale of Perceived Social Support, Kessler Psychological Distress Scale and Health Services Utilization questionnaires (for indirect costs), and compared between HD and PD patients.

Results from this study will provide important HRQoL information to assist renal physicians and patients to make treatment decisions. Furthermore, intervention programs could be developed to improve social support based on patients' needs. These could in turn improve patients' HRQoL, morbidity and mortality outcomes with minimal risks involved.

ELIGIBILITY:
Inclusion Criteria:

* All chronic HD and PD patients who are on regular follow-up with nephrologists in the NUH outpatient renal or PD clinic, and who meet the following criteria will be included in the study: male or female 21 years of age or older, with stage 5 CKD (eGFR <15 ml/min/1.73m2) and have been receiving HD or PD for at least 3 months.

Exclusion Criteria:

* Transient dialysis patients, those have poor cognitive function or are not able to complete the questionnaires or give informed consent.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stage 5 chronic kidney disease hemodialysis peritoneal dialysis
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2012-01; Primary Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Patient-Reported, Economic and Clinical Outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Priscilla P How, Pharm.D., Principal Investigator — National University of Singapore
Locations (1):
- National University of Singapore, Singapore, Singapore, Singapore